CLINICAL TRIAL: NCT00503490
Title: Phase I, Single and Multi-dose, Placebo Controlled, Randomized, Dose-Escalation Study to Evaluate the Safety, Tolerability and PK Profile of MP-376 Using the PARI eFlow Nebulizer for 14 Days to CF Patients
Brief Title: Safety, Pharmacokinetic and Pharmacodynamic Study of MP-376 in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mpex-203
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Inhaled Levofloxacin
  Interventions: Drug: MP-376 (Levofloxacin solution for Inhalation)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MP-376 (Levofloxacin solution for Inhalation) — 40, 80, 120mg RDD
  Arms: 1
Drug: placebo — BID
  Arms: 2

SUMMARY:
Patients with cystic fibrosis (CF) suffer from chronic infections of the lower respiratory tract that can be caused by one or multiple bacteria, including Pseudomonas aeruginosa, which has been particularly problematic to eradicate and been implicated as the major cause of morbidity and mortality in CF patients. Aerosol delivery of antibiotics directly to the lung increases the local concentrations of antibiotic at the site of infection resulting in improved antimicrobial effects compared to systemic administration. Bacterial resistance to current aerosol antibiotic treatments indicate a need for improved therapies to treat CF patients with pulmonary infections caused by multi-drug resistant Pseudomonas aeruginosa and other bacteria. High concentrations of MP-376 delivered directly to the lung are projected to have antimicrobial effects on even the most resistant organisms and reduce the emergence of resistant bacteria.

DETAILED DESCRIPTION:
This trial will be a single-blind, placebo-controlled, dose escalating between cohorts, single and multi-dose, multi-center study to evaluate the safety, tolerability and pharmacokinetic profile of levofloxacin administered as MP-376 once, then twice daily for 14 days by the aerosol route to CF patients.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* > 16 years of age
* Confirmed Diagnosis of Cystic Fibrosis
* Positive sputum culture for P. aeruginosa within the past 6 months
* Patients are able to elicit an FEV1 >/= 40% of predicted value at screening
* Clinically stable with no evidence of acute respiratory or lower respiratory infections within 28 days prior to dosing
* Able to reproducibly perform spirometry measurements and be able to repeatedly produce sputum over several hours

Exclusion Criteria:

* Use of any nebulized or systemic antibiotics within 4 weeks of starting study
* History of hypersensitivity to fluoroquinolones or intolerance with aerosol medication
* Uncontrolled diabetes or abnormal renal function
* Tobacco use (smoking) in the last 30 days

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MP-376 administered twice a day for 14 days | 14 days

SECONDARY OUTCOMES:
Evaluate changes in the microbiology of CF sputum after 14 days of treatment with MP-376 | 14 days
PK Profile of single-dose vs multi-dose of MP-376 | 14 days
Evaluate changes in FEV1 and FVC over 14 days of Treatment | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (13):
- United States (13):
  - La Jolla, California
  - Los Angeles, California
  - Palo Alto, California
  - Orlando, Florida
  - Kalamazoo, Michigan
  - Omaha, Nebraska
  - Albany, New York
  - New Hyde Park, New York
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Charleston, South Carolina
  - San Antonio, Texas
  - Salt Lake City, Utah